CLINICAL TRIAL: NCT05828550
Title: Detection of Efflux Pump Genes Mediating Ciprofloxacin Resistance in Staphylococcus Aureus Isolates in Sohag University Hospitals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Esaam Eldin Farrag, demonestrator at microbiology and Immunology department, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-04-01MS
Record Dates: First submitted 2023-04-13; First posted 2023-04-25 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Patients withInfections Caused by S.Aureus Like Skin Infections , Chest Infections , Surgical Site Infections , and Urinary Tract Infections
MeSH Terms: conditions — Surgical Wound Infection; Urinary Tract Infections | interventions — Drug Collateral Sensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: antibiotic sensitivity — The resistance pattern of the isolates will be detected by disc diffusion method.
  Detection of efflux pump genes responsible for the resistance ( norA , norB , norC ) by PCR
  Other Names: polymerase chain reaction

SUMMARY:
Among multidrug-resistant bacteria, Methicillin-resistant Staphylococcus aureus (MRSA) isolates were recognized to be an important mortality factor in hospital infections and a major concern in health-care and community settings . The antibiotic-resistant of S. aureus is extended by various bacterial strategies, including limiting uptake of the drug, alteration of the drugtargets, production of druginactivating enzymes and the activation of efflux pumps that effectively remove antibiotics . Relying on the type of antibiotics, bacteria can apply one or more strategies. Specifically, localization of resistance genes in transferable genetic elements, such as plasmid and transposons , causing Horizontal transfer of resistance genes between bacterial strains . MRSA strains are resistant to nearly all beta-lactam antibiotics by producing an alternative penicillin-binding protein known as PBP2a . This protein is encoded by the mecA gene and has a low affinity to manybeta-lactam antibiotics. Furthermore, these strains often show resistance to a wide range of antibiotics . The use of fluoroquinolone for the effective infectious therapy is limited by presence of fluoroquinolone resistance . There are two mechanisms causing resistance to fluoroquinolone. The first one is attributed to mutations occurring in the quinolone-resistance determining region (QRDR) of topoisomerase IV encoded by grlA/grlB and DNA gyrase encoded by gyrA/gyrB; these mutations decrease the affinity ofthe drug. The other mechanism is mediated by efflux pumps which is less recognized . Recently, several efflux pumps have been identified for S. aureus including efflux pumps encoded by chromosome or plasmids. The efflux pumps norA, norB, norC, mdeA, sepA, mepA, sdrM and lmrS are encoded by chromosome while qacA/B, qacG, qacH, qacJ and smr are plasmid-encoded . Efflux pumps could be specialized for specific substrate or mobilized a wide varieties of different antibiotic classes . Despite, efflux pumps can potentially increase resistance to antibiotics in clinical isolates of S. aureus, few studies have been evaluated the individual and collective participation of the efflux system in resistant isolates . Therefore the aim of the study is to detect ciprofloxacin resistant strains of staphylococcus aureus isolates and to detect efflux pump genes ( norA , norB and norC ) mediating resistance in such strains.

ELIGIBILITY:
Inclusion Criteria:

* Infections caused by S.aureus like skin infections , chest infections , surgical site infections , and urinary tract Infections

Exclusion Criteria:

* Infections caused by any organisms other than S.aureus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Ciprofloxacin Resistance in Staphylococcal strains isolated | 6 months
  resistance pattern of the isolates will be detected by disc diffusion method
presence of Efflux pump genes ( norA , norB , norC ) mediating Resistance in such strains | 6 months
  Detection of efflux pump genes responsible for the resistance ( norA , norB , norC ) by PCR

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Havaei S, Moghadam SO, Pourmand M, Faghri J. Prevalence of Genes Encoding Bi-Component Leukocidins among Clinical Isolates of Methicillin Resistant Staphylococcus aureus. Iran J Public Health. 2010;39(1):8-14. Epub 2010 Mar 31. PMID 23112984
- [Background] Lowy FD. Antimicrobial resistance: the example of Staphylococcus aureus. J Clin Invest. 2003 May;111(9):1265-73. doi: 10.1172/JCI18535. No abstract available. PMID 12727914
- [Background] Pourmand MR, Yousefi M, Salami SA, Amini M. Evaluation of expression of NorA efflux pump in ciprofloxacin resistant Staphylococcus aureus against hexahydroquinoline derivative by real-time PCR. Acta Med Iran. 2014;52(6):424-9. PMID 25130148
- [Background] Yilmaz ES, Aslantas O. Antimicrobial resistance and underlying mechanisms in Staphylococcus aureus isolates. Asian Pac J Trop Med. 2017 Nov;10(11):1059-1064. doi: 10.1016/j.apjtm.2017.10.003. Epub 2017 Nov 8. PMID 29203102